CLINICAL TRIAL: NCT02915510
Title: Evaluating the Tolerance, Safety and Acceptability of PKU GMPro, a Whey Protein Derived Feed for the Dietary Management of Phenylketonuria in Children and Adults - a Pilot Trial
Brief Title: GMP Drink for PKU Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nutricia UK Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: GMP2016
Record Dates: First submitted 2016-08-08; First posted 2016-09-27 (Estimated); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Phenylketonuria
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GMP (Experimental): Single arm designed, 3 day baseline, 28day on GMP
  Interventions: Dietary Supplement: Glycomacropeptide-based protein substitute

INTERVENTIONS:
Dietary Supplement: Glycomacropeptide-based protein substitute

SUMMARY:
This study will evaluate the safety, gastrointestinal (GI) tolerance, acceptability and compliance of a Glycomacropeptide-based protein substitute for patients with Phenylketonuria (PKU).

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Over 3 years of age
* Diagnosed with classical or variant type phenylketonuria
* Have been compliant in taking at least one amino acid-based, Phe-free protein substitute, providing at least 20g protein equivalents, for at least 1 month prior to trial commencement
* Have a prescribed daily Phe allowance
* Written informed consent from patient, or from parent / carer if applicable

Exclusion Criteria:

* Currently prescribed Sapropterin or similar tetrahydrobiopterin based medication
* Pregnant or lactating
* Requiring parenteral nutrition
* Major hepatic or renal dysfunction
* Participation in other studies within 1 month prior to entry of this study
* Allergy to any of the study product ingredients, including milk protein or soya
* Investigator concern around willingness/ability of patient or parent/carer to comply with protocol requirements

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-07; Primary Completion 2019-09-27 (Actual); Study Completion 2019-09-27 (Actual)

PRIMARY OUTCOMES:
Blood Phenylalanine (and other amino acids) | 3 points throughout 28 days
  Blood spot test

SECONDARY OUTCOMES:
Gastro-intestinal tolerance questionaire | 12/31 days
  Questionaire detailing any GI symptoms, severity and change from usual
Product compliance questionaire | 31 days
  Breif questionaire on amounts offered and amounts actually consumed, compared to recomended amount.
Product acceptability questionnaire | 2/31 days
  Breif tick-box questionaire on overal liking and acceptability of product
Patient reproted nutrient intake (3 day food diaries) | 6/31 days
  3 day food diaries, subsequently analysed in dietary software.
Pateint-reported appetite (visual analogue scale) | 6/31 days
  Measures of overal appetite and satiety via visual analouge scale
Antropometry (hieight and weight) | 2/31 days
  Measurements of height and weight at baseline and end of study
Safety (Adverse events reporting) | 31 days
  Reporting of adverse events throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Stratton, PHd, Study Director — Nutricia Ltd UK
Locations (5):
- United Kingdom (5):
  - Great Ormond Street Hospital, London
  - Guy's and St Thomas' NHS Fondation Trust, London
  - UCLH, London
  - Royal Manchester Children's Hospital, Manchester
  - Sheffield Teaching Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: No